CLINICAL TRIAL: NCT03879993
Title: Effects of Resistance Training in People Living With HIV/AIDS
Brief Title: Resistance Training in People Living With HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of Maringá (Other)
Responsible Party: Principal Investigator, Ademar Avelar de Almeida Junior, Principal Investigator, State University of Maringá
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Exercise and HIV
Record Dates: First submitted 2019-03-12; First posted 2019-03-19 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: HIV/AIDS
Keywords: Exercise; Cognition; Body composition; Inflammatory biomarkers; CD4
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blood collections and subsequent analyzes were done blindly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Exercise group was resistance training three times per week, during 45 to 60 minutes per day. Training program was composed by bench press, leg press 45°, lat pulldown, knee extension, dumbbell lateral raise, horizontal leg curl, triceps pulldown, seated calf raise, biceps curls and abdominal. Participants should complete 3 series with 8-12 repetitions of each exercise, which was supervised by trained research personnel. There were 60 seconds of interval between series and exercises were separated by a 120 seconds recovery period.
  Interventions: Other: Exercise group
- Control group (No Intervention): Control group was not do any exercise during intervention period. Participants was asked to keep their habitual routine until finish the final evaluations.

INTERVENTIONS:
Other: Exercise group — Resistance training 3 times per week (45-60 minutes of resistance training)
  Other Names: Training group
  Arms: Exercise group

SUMMARY:
The aim of this study will be to verify effects of resistance training in people living with HIV/AIDS.

DETAILED DESCRIPTION:
The aim of this study was verify effects of resistance training in cognitive function, body composition and biochemical parameters of inflammation and oxidative stress in people living with HIV/AIDS. The sample was composed by patients with HIV/AIDS of both sexes. The patients were randomized in two groups, a exercise group (EG), which was receive intervention with eight weeks of resistance training, and a control group (CG), that was not to do exercise. The cognitive function was analyzed with Stroop Test and Trail Test; body composition was evaluated by bioimpedance; blood tests was use to analyze biochemical parameters of inflammation and oxidative stress. For statistical analysis was used ANOVA of two factors for repeated measurements, having the (EG and PG) group and the time (pre and post exercise). Level of significance adopted was P < 0,05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnostic for HIV/AIDS.
* Clinical condition and viral count stabilized.
* Have been using (HAART) for 6 months or more.
* Not have participated in physical exercise programs in six months before beginning of study.
* Not have muscle or joint injuries that make it impossible to practice physical activity.
* Not be pregnant.

Exclusion Criteria:

* Not attending more than 15% of the intervention sessions or visits to the laboratory.
* Aggravation of the disease.
* Stick to a physical activity program in addition to that offered by the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Cognitive Function | Baseline and eight weeks
  Victoria Stroop, Castro Cunha & Martins Stroop and Trail Test were performed at baseline and after eight weeks of intervention in both groups (EG and CG). Blood will be collected and brain-derived neurotrophic factor (BDNF) will be measured by Enzyme-Linked Immunosorbent Assay Method (Human - ELISA Kit) at baseline and after eight weeks of intervention in both groups (EG and CG).

SECONDARY OUTCOMES:
CD4 / CD8 | Baseline and eight weeks
  Blood was collected and cluster of differentiation 4 (T CD4+) and cluster of differentiation 8 (T CD8+) cells was measured by flow cytometry (BD TrucountTM Tubes) with FACSCalibur (Dickinson, New Jersey, USA) at baseline and after eight weeks of intervention in both groups (EG and CG).
Concentration of Inflammatory markers | Baseline and eight weeks
  Blood was collected and interferon (INF-y), interleukin 4 (IL-4), interleukin 6 (IL-6) and interleukin 10 (IL-10) was be measured by Enzyme-Linked Immunosorbent Assay Method (Human - ELISA Kit) at baseline and after eight weeks of intervention in both groups (EG and CG).
Health cellular | Baseline and eight weeks
  Cellular health was evaluated through phase angle value using the bio-electrical bioimpedance method (Biodynamics 450 analyzer, Biodynamics Corporation, Seattle, USA) at baseline and after eight weeks of intervention in both groups (EG and CG).

OTHER OUTCOMES:
Change in body composition | Baseline and eight weeks
  Body composition was evaluated at baseline and after eight weeks of intervention in both groups (EG and CG) using thickness of skin folds (Lange Adipometer). The skin folds of the triceps, subscapular, supra iliac, abdominal, thigh and leg were collected. The data were inserted into formulas appropriate to the population studied for calculating body composition.
Change in body circumferences | Baseline and eight weeks
  Perimeters of arms, chest, abdomen, waist, hip, thigh and leg were measured at baseline and after eight weeks of intervention in both groups (EG and CG).
Change brachial blood pressure | Baseline and eight weeks
  Brachial blood pressure (systolic and diastolic pressures) was assessed through an automatic monitor (HEM-742, Omron Healthcare, Japan) at baseline and after eight weeks of intervention in both groups (EG and CG).
Change autonomic cardiac modulation | Baseline and eight weeks
  The autonomic cardiac modulation was evaluated through a heart rate monitor (Polar, model RS-800, USA) at baseline and after eight weeks of intervention in both groups (EG and CG).
Change in handgrip strength | Baseline and eight weeks
  Handgrip strength was evaluated by handgrip dynamometer at baseline and after eight weeks of intervention in both groups (EG and CG).
Change in flexibility | Baseline and eight weeks
  Flexibility was evaluated by sit and reach test at baseline and after eight weeks of intervention in both groups (EG and CG).
Training load control | Baseline and eight weeks
  Training load control was done by weekly monitoring and adjustment of the weights (kg) used in each exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Ademar Avelar, PhD, Principal Investigator — State University of Maringá
Locations (1):
- State University of Maringá, Maringá, Paraná, Brazil

REFERENCES:
- [Background] de Assis GG, de Almondes KM. Exercise-dependent BDNF as a Modulatory Factor for the Executive Processing of Individuals in Course of Cognitive Decline. A Systematic Review. Front Psychol. 2017 Apr 19;8:584. doi: 10.3389/fpsyg.2017.00584. eCollection 2017. PMID 28469588
- [Background] Di Benedetto S, Muller L, Wenger E, Duzel S, Pawelec G. Contribution of neuroinflammation and immunity to brain aging and the mitigating effects of physical and cognitive interventions. Neurosci Biobehav Rev. 2017 Apr;75:114-128. doi: 10.1016/j.neubiorev.2017.01.044. Epub 2017 Feb 1. PMID 28161508
- [Background] Bossers WJ, van der Woude LH, Boersma F, Hortobagyi T, Scherder EJ, van Heuvelen MJ. A 9-Week Aerobic and Strength Training Program Improves Cognitive and Motor Function in Patients with Dementia: A Randomized, Controlled Trial. Am J Geriatr Psychiatry. 2015 Nov;23(11):1106-16. doi: 10.1016/j.jagp.2014.12.191. Epub 2015 Jan 3. PMID 25648055
- [Background] Dinoff A, Herrmann N, Swardfager W, Lanctot KL. The effect of acute exercise on blood concentrations of brain-derived neurotrophic factor in healthy adults: a meta-analysis. Eur J Neurosci. 2017 Jul;46(1):1635-1646. doi: 10.1111/ejn.13603. Epub 2017 Jun 19. PMID 28493624
- [Background] Dufour CA, Marquine MJ, Fazeli PL, Henry BL, Ellis RJ, Grant I, Moore DJ; HNRP Group. Physical exercise is associated with less neurocognitive impairment among HIV-infected adults. J Neurovirol. 2013 Oct;19(5):410-7. doi: 10.1007/s13365-013-0184-8. Epub 2013 Aug 10. PMID 23934585
- [Background] Fazeli PL, Woods SP, Heaton RK, Umlauf A, Gouaux B, Rosario D, Moore RC, Grant I, Moore DJ; HNRP Group. An active lifestyle is associated with better neurocognitive functioning in adults living with HIV infection. J Neurovirol. 2014 Jun;20(3):233-42. doi: 10.1007/s13365-014-0240-z. Epub 2014 Feb 20. PMID 24554483
- [Background] Ghafouri M, Amini S, Khalili K, Sawaya BE. HIV-1 associated dementia: symptoms and causes. Retrovirology. 2006 May 19;3:28. doi: 10.1186/1742-4690-3-28. PMID 16712719
- [Background] McDermott A, Zaporojan L, McNamara P, Doherty CP, Redmond J, Forde C, Gormley J, Egana M, Bergin C. The effects of a 16-week aerobic exercise programme on cognitive function in people living with HIV. AIDS Care. 2017 Jun;29(6):667-674. doi: 10.1080/09540121.2016.1263723. Epub 2016 Nov 28. PMID 27892704
- [Background] de Souza DC, da Silva JC, Matos FO, Okano AH, Bazotte RB, Avelar A. The Effect of a Short Period of Supplementation with Glutamine Dipeptide on the Cognitive Responses after a Resistance Training Session of Women with HIV/AIDS: A Randomized Double-Blind Placebo-Controlled Crossover Study. Biomed Res Int. 2018 Apr 3;2018:2525670. doi: 10.1155/2018/2525670. eCollection 2018. PMID 29850491
- [Background] Llames L, Baldomero V, Iglesias ML, Rodota LP. [Values of the phase angle by bioelectrical impedance; nutritional status and prognostic value]. Nutr Hosp. 2013 Mar-Apr;28(2):286-95. doi: 10.3305/nh.2013.28.2.6306. Spanish. PMID 23822677
- [Background] Meynell J, Barroso J. Bioimpedance analysis and HIV-related fatigue. J Assoc Nurses AIDS Care. 2005 Mar-Apr;16(2):13-22. doi: 10.1016/j.jana.2005.01.006. PMID 16438122
- [Background] Gupta D, Lammersfeld CA, Burrows JL, Dahlk SL, Vashi PG, Grutsch JF, Hoffman S, Lis CG. Bioelectrical impedance phase angle in clinical practice: implications for prognosis in advanced colorectal cancer. Am J Clin Nutr. 2004 Dec;80(6):1634-8. doi: 10.1093/ajcn/80.6.1634. PMID 15585779
- [Background] Schwenk A, Beisenherz A, Romer K, Kremer G, Salzberger B, Elia M. Phase angle from bioelectrical impedance analysis remains an independent predictive marker in HIV-infected patients in the era of highly active antiretroviral treatment. Am J Clin Nutr. 2000 Aug;72(2):496-501. doi: 10.1093/ajcn/72.2.496. PMID 10919947
- [Background] Ott M, Fischer H, Polat H, Helm EB, Frenz M, Caspary WF, Lembcke B. Bioelectrical impedance analysis as a predictor of survival in patients with human immunodeficiency virus infection. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 May 1;9(1):20-5. PMID 7712230
- [Background] Tomeleri CM, Ribeiro AS, Cavaglieri CR, Deminice R, Schoenfeld BJ, Schiavoni D, Dos Santos L, de Souza MF, Antunes M, Venturini D, Barbosa DS, Sardinha LB, Cyrino ES. Correlations between resistance training-induced changes on phase angle and biochemical markers in older women. Scand J Med Sci Sports. 2018 Oct;28(10):2173-2182. doi: 10.1111/sms.13232. Epub 2018 Jun 25. PMID 29858504
- [Background] Souza MF, Tomeleri CM, Ribeiro AS, Schoenfeld BJ, Silva AM, Sardinha LB, Cyrino ES. Effect of resistance training on phase angle in older women: A randomized controlled trial. Scand J Med Sci Sports. 2017 Nov;27(11):1308-1316. doi: 10.1111/sms.12745. Epub 2016 Aug 19. PMID 27541287
- [Background] Deresz LF, Scholer CM, de Bittencourt PIHJ, Karsten M, Ikeda MLR, Sonza A, Dal Lago P. Exercise training reduces oxidative stress in people living with HIV/AIDS: a pilot study. HIV Clin Trials. 2018 Aug;19(4):152-157. doi: 10.1080/15284336.2018.1481247. Epub 2018 Oct 27. PMID 30369300
- [Derived] de Souza DC, Marchini KB, Nunhes PM, Domingues WJR, Bertolini DA, Oliveira V, Mazzardo O, Avelar A. Resistance Training Improves Cognitive Function and Depression Without Changing BDNF Levels in People Living with HIV: a Randomized Controlled Clinical Trial. AIDS Behav. 2025 Dec;29(12):3877-3886. doi: 10.1007/s10461-025-04824-6. Epub 2025 Jul 25. PMID 40711680